CLINICAL TRIAL: NCT03033524
Title: A Multicenter, 3-Arm, Open-Label, Phase Ⅱa Clinical Trial to Evaluate the Safety and Efficacy of TTAC-0001, a Fully Human Monoclonal Antibody in Patients With Recurrent Glioblastoma
Brief Title: Trial to Evaluate the Safety of TTAC-0001(Tanibirumab) in Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmAbcine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMC_TTAC-0001_02
Record Dates: First submitted 2017-01-09; First posted 2017-01-26 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — olinvacimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Patients will be treated with 8mg/kg of TTAC-0001 on day 1, day 8 and day 15 in every 4 weeks of cycle.
  Interventions: Drug: TTAC-0001
- Cohort 2 (Experimental): Patients will be treated with 12mg/kg of TTAC-0001 on day 1, day 8 and day 15 in every 4 weeks of cycle.
  Interventions: Drug: TTAC-0001
- Cohort 3 (Experimental): Patients will be treated with 12mg/kg of TTAC-0001 weekly in every 4 weeks of cycle.
  Interventions: Drug: TTAC-0001

INTERVENTIONS:
Drug: TTAC-0001 — Calculated amount of drug will be diluted with normal saline and administered intravenously.
  Other Names: Tanibirumab

SUMMARY:
Study Design - Multicenter, open-label, 3 arms, stepwise, phase Ⅱa clinical trial

Study objective:

1. Primary - To evaluate the safety of TTAC-0001 in patients with recurrent glioblastoma.
2. Secondary - To determine the efficacy of TTAC-0001 in patients with recurrent glioblastoma.
3. Exploratory

   * To evaluate pharmacokinetic (PK) parameters of TTAC-0001 in patients with recurrent glioblastoma
   * To evaluate pharmacodynamic (PD) parameters by clinical biomarker test

Study Methodology

Patients will be sequentially enrolled from the 1st arm. An enrollment criterion to the next arm is defined as no patients in the previous treatment arm showing grade ≥3 of hemangioma or other Dose Limiting Toxicities (DLT). A safety review committee (SRC) will convene to determine the patient's safety with a decision on enrollment into the next arm or change in dosing frequency of study drug in the above case.

A patient who is withdrawn from the study before the completion of the 1st cycle can be replaced with another patient. Patients will be treated for up to 1 year, unless a cause for termination occurs, such as progression of disease (PD) or the withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients ≥19 years old
* Diagnosed with primary glioblastoma by histopathological examination and confirmed recurrent glioblastoma by magnetic resonance imaging (MRI) scans after concomitant temozolomide chemotherapy with radiotherapy (CCRT). One previous recurrence/progression of glioblastoma with reintroduction/altered schedule of temozolomide is allowable.
* At least one confirmed measurable lesion or non measurable lesion by response assessment in neuro-oncology (RANO) criteria
* Karnofsky Performance Status (KPS) ≥ 80
* A person who satisfies the following criteria in hematologic, renal, and hepatic function tests
* At least 12 weeks of expected survival time
* Signed informed consent

Exclusion Criteria:

* Diagnosed with other malignant tumor within 2years
* Uncontrolled HT or seizure, class III or IV heart failure, oxygen dependent disease, active psychiatric disorder
* Not recovered grade 2 AE due to previous CCRT
* Major surgery or other investigational drug treatment within 4 weeks
* Pregnant/lactating female and female/male potential childbearing without contraception
* Severe drug hypersensitivity or hypersensitivity to a therapy similar to the study drug
* Expectation of poor compliance
* Previous therapy with VEGF targeted agent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | up to 1 year

SECONDARY OUTCOMES:
PFS at 6-month time point | 6 months
Objective response rate (ORR) | up to 1 year
  The rate of complete response and partial response assessed according to RANO criteria.
Disease control rate(DCR) | up to 1 year
  The rate of complete response(CR), partial response(PR) and stable disease(SD) assessed according to RANO criteria.
Overall survival(OS) | up to 1 year

OTHER OUTCOMES:
Area under the concentration-time curve (AUC) | up to 1 year
  Pharmacokinetics profile
Maximum plasma concentration (Cmax) | up to 1 year
  Pharmacokinetics profile
Minimum plasma concentration (Cmin) | up to 1 year
  Pharmacokinetics profile
Clearance (CL) | up to 1 year
  Pharmacokinetics profile
Volume of distribution (Vd) | up to 1 year
  Pharmacokinetics profile
Half-life (t1/2) | up to 1 year
  Pharmacokinetics profile
Angiogenic factors in serum or changes in concentration | up to 1 year
  Pharmacodynamics profile
Perfusion parameter assessed by DCE-MRI | every 2 cycles(each cycle is 4 weeks), up to 1year
  Pharmacodynamics profile
Expression of angiogenic factors in endothelial cells | At screening
  Analyzed by IHC of tumor tissue
Immunogenicity | Day 1 of every cycle(each cycle is 4 weeks), up to 1 year
  Anti-drug (TTAC-0001) antibody (ADA) test for evaluation of immunogenicity

IPD SHARING:
Plan to Share IPD: Undecided